CLINICAL TRIAL: NCT04749225
Title: Assessment of a Properly Video Stylet Angulation for Nasotracheal Intubation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pin-Yang Hu, MD, Physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUHIRB-F(I)-20200202
Record Dates: First submitted 2021-02-02; First posted 2021-02-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Intubation Complication
Keywords: video stylet; angulation; nasotracheal intubation; trachway; tracheal intubation; Endotracheal Tube intubation General Anesthesia (ETGA)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — *undergoing oro-maxillofacial surgery with general anesthesia(GA) *ASA(American Society of Anesthesiologists):Ι to III -20 to 65 years old *mouth open > 3cm *the systemic disease exclusion/conscious clear and without major Neurocognitive Disorder
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 45° group: Uses the video stylet with 45 degree(The tip of the trachway in 45°-55°) to assist the nasotracheal tube passing the nasal cavity, oropharynx and advanced into the trachea
- 70° group: Uses the video stylet with 70 degree(The tip of the trachway in 60°-70°)to assist the nasotracheal tube passing the nasal cavity, oropharynx and advanced into the trachea
- 90° group: Uses the video stylet with 90 degree(The tip of the trachway in 80°-90°)to assist the nasotracheal tube passing the nasal cavity, oropharynx and advanced into the trachea

SUMMARY:
Uses the video stylet with different angulation to assist the nasotracheal tube passing the nasal cavity, oropharynx and advanced into the trachea.

DETAILED DESCRIPTION:
In oro-maxillo-facial surgery, it is a common practice for patients receiving general anesthesia with nasotracheal intubation to widen the surgical field and to ease undergoing surgery. However, a nasotracheal tube blindly passing through the nasal cavity may easily result in nasal cavity and oropharynx damages.

The aim of the study is to investigate use which angulation including 45 degree, 70 degree and 90 degree is appropriate to assist the nasotracheal tube passing the nasal cavity, oropharynx, and advanced into the tracheal. Patients are randomized into three groups by 45 degree, 70 degree and 90 degree to facilitate nasotracheal tube sliding through into trachea and compared with each other group.

Hemodynamic changes in each time interval, each time taken of tube going through the nasal cavity, tube advanced from oropharynx into trachea will be recorded. The incidence of using the video stylet with different angulation to accurately place tube tip into trachea, intubation related side effects and complications are recorded at postoperative time stages.

ELIGIBILITY:
Inclusion Criteria:

* undergoing oro-maxillofacial surgery with general anesthesia(GA)
* ASA(American Society of Anesthesiologists):Ι to III
* 20-65 y/o
* mouth Open > 3cm
* the systemic disease exclusion
* conscious clear and without major Neurocognitive Disorder
* Mandarin or Taiwanese speaker
* agree the purpose of the study and sign the ICF

Exclusion Criteria:

* difficult airway assessment [limited mouth opening<3cm, limited neck motion(thyromental distance < 6cm]
* previous head neck surgery history
* upper abnormal airway diagnosed, easily epistaxis, and both sides nasal cavities obstruction.
* reject to participate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult(20-65 years old)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
success rate of video stylet angulation and successful first tube attempt in 60 seconds | During procedure
  Time: TTI(time taken advancement) is less than 60 seconds in first tube attempt, it defines successful; TTI(time taken advancement) is over 60 seconds in first tube attempt, it defines unsuccessful.
success rate of video stylet angulation and successful first tube attempt in Lung's ventilation | During procedure
  Lung's ventilation: The lung's ventilation is success.
time taken advancement(TTI) | During procedure
  time taken advancement from nasal cavity into trachea in each time interval
assessment of difficult intubation(IDS) | During procedure
  Assessment of difficult intubation by Intubation Difficulty Scale(The Intubation Difficulty Scale, IDS, 1997) is required after intubation. Number of Attempts>1, score "N1"; Number of Operators >1, score "N2"; Number of Alternative Techniques, score "N3"; Comark Grade -1, score "N4"; Lifting Force Required Normal, score "N5=0"; Lifting Force Required Increased, score "N5=1"; Laryngeal Pressure Not applied, score "N6=0"; Laryngeal Pressure Applied, score "N6=1"; Vocal Cord Mobility Abducion, score "N7=0"; Vocal Cord Mobility Adducion, score "N7=1". IDS=Sum of scores(N1-N7). If IDS score gains "0" means "Easy", "0<IDS≤5" means "Slight Difficulty", "5<IDS" means "Moderate to Major Difficulty", "IDS=∞" means "Impossible intubation".
assessment of Glottic grade(Cormack Grade) | During procedure
  Assessment of Glottic grade(Cormack Grade) is required after intubation. The definitions of grade: Grade 1: full view of the glottis; Grade 2a: partial view of the glottis; Grade 2b: arytenoids only; Grade 3: epiglottis only; Grade 4: neither glottis or epiglottis identified

SECONDARY OUTCOMES:
post-intubation induced oropharyngeal bleeding, hoarseness and sore throat | Day 2(the day after the operation)
  A visiting questionnaire is used to measure the condition of post-intubation, including oropharyngeal bleeding, sore throat, hoarseness, dysphagia. The score for the measurement of oropharyngeal bleeding, sore throat, hoarseness, dysphagia is divided into four degrees: none, mild, moderate and severe. All the evaluation will be assessed in the next coming morning after the postoperation.

CONTACTS AND LOCATIONS:
Overall Officials: Pin-Yang Hu, MD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin District, Taiwan